CLINICAL TRIAL: NCT07103486
Title: Retrospective Chart Review for German Adult Patients With Relapsed or Refractory Diffuse Large B-cell Lymphoma (DLBCL) After Two or More Lines of Systemic Therapy With Subsequent Historical Comparison Against Tisagenlecleucel Based on JULIET Trial (CTL019C2201)
Brief Title: A Study to Evaluate the Therapeutic Benefit of Tisagenlecleucel Compared to Existing Standard of Care in German Adult Patients With Relapsed or Refractory Diffuse Large B-cell Lymphoma
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CCTL019CDE01
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: Relapsed; Refractory
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- Tisagenlecleucel Full Analysis Set (FAS) Group: Adult patients with r/r DLBCL who were enrolled in the JULIET trial and received an infusion of tisagenlecleucel.
- Tisagenlecleucel Intention To Treat (ITT) Group: Adult patients with r/r DLBCL who were enrolled in the JULIET trial.
- External Control Group: Adult patients with r/r DLBCL after two or more lines of chemotherapy. Patient data was collected from German medical center chart reviews.

SUMMARY:
The aim of this study was to evaluate the therapeutic benefit of tisagenlecleucel compared to the existing standard of care in adult patients with relapsed or refractory diffuse large B-cell lymphoma (r/r DLBCL). For tisagenlecleucel patients, patient-level data from the JULIET study (CTL019C2201) was used. Data for patients treated with the appropriate comparator therapy (ACT) in German routine care was collected via chart review by 8 medical centers in Germany. The medical charts provided data on adult patients at the time of the qualifying treatments in the time period from approximately 2010 to 2017 with the longest possible follow-up phases (up to 5 years, but only until December 31, 2020).

ELIGIBILITY:
Inclusion criteria:

* Aged 18 years or older.
* Histologically confirmed DLBCL, transformed indolent Non-Hodgkin Lymphoma (NHL) was also allowed (such as transformed follicular lymphoma).
* r/r DLBCL after 2 or more chemotherapy lines, including rituximab and anthracycline. Previous autologous hematopoietic stem cell transplantation (HSCT) was allowed. For transformed indolent NHL, anthracycline treatment before transformation was allowed.
* Had received patient-individual therapy in the qualifying line(s) (3rd or to a maximum of 9th line). Patient-individual therapy was chosen in consideration of molecular genetic lymphoma characteristics, previous therapies, disease history and patient's general condition, including an allogeneic HSCT where possible. Best supportive care in the palliative setting was also a treatment option.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. Even if no ECOG performance status or Karnofsky Index was documented in patient charts the patient could be eligible for documentation.
* Had adequate organ function at the discretion of the treating physician:

  * Adequate pulmonary reserve (e.g. ≤ Grade 1 dyspnea and pulse oxygenation > 91 % on room air)
  * Hemodynamically stable and adequate cardiac function (e.g. Left Ventricular Ejection Fraction (LVEF) ≥ 45 %)

Exclusion criteria:

* Received more than 8 treatment lines before qualifying treatment failure.
* Active central nervous system (CNS) involvement by malignancy.
* Had prior allogeneic HSCT.
* Human immunodeficiency virus (HIV)-positive patients.
* Had uncontrolled, acutely life-threatening bacterial, viral or mycotic infections (e.g. blood culture positive ≤ 72 hours before treatment start).
* Had unstable angina pectoris and/or myocardial infarct within 6 months before qualifying treatment failure.
* Had previous or concurrent malignant tumor disease with some exceptions (basal cell or squamous cell carcinoma, curatively treated in-situ carcinoma of the cervix or breast, curatively treated primary malignant tumor disease in complete remission for ≥ 5 years).
* Had cardiac arrhythmias that could not be controlled with drug treatment.
* Patients with T-cell-rich/histiocyte-rich large B-cell lymphoma (THRBCL), primary cutaneous large B-cell lymphoma, primary mediastinal B-cell lymphoma (PMBCL), Epstein Barr virus (EBV)-positive DLBCL in the elderly, Richter's transformation, and Burkitt lymphoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 264 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to approximately 5 years
  For the external control and tisagenelcleucel FAS groups: OS was defined as the time from the date of treatment start to the date of death due to any cause and censored otherwise.
  For the tisagenelcleucel ITT group: OS was defined as the time from the date of enrollment to the date of death due to any cause and censored otherwise.
Progression-free Survival (PFS) | Up to approximately 5 years
  For the external control and tisagenelcleucel FAS groups: PFS was defined as the time from the date of treatment start to the date of first documented disease progression or death due to any cause and censored otherwise.
  For the tisagenelcleucel ITT group: PFS was defined as the time from the date of enrollment to the date of first documented disease progression or death due to any cause and censored otherwise.
Event-free Survival (EFS) | Up to approximately 5 years
  For the external control and tisagenelcleucel FAS groups: EFS was defined as the time from the date of treatment start to the date of first documented disease progression or relapse, new treatment for lymphoma or death due to any cause and censored otherwise.
  For the tisagenelcleucel ITT group: EFS was defined as the time from the date of enrollment to the date of first documented disease progression or relapse, new treatment for lymphoma or death due to any cause.
Overall Response Rate (ORR) | Up to approximately 5 years
  ORR was defined as the proportion of patients with a best overall disease response of complete response (CR) or partial response (PR), respectively until progressive disease or start of new anticancer therapy, whichever came first. CR and PR efficacy evaluation was based on Cheson Response Criteria and The Lugano Classification (2014).

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States